CLINICAL TRIAL: NCT07271888
Title: Effect of Mendelsohn Maneuver, Effortful Swallow Training, and the Shaker Exercise on Swallowing Ability Among Dysphagic Patients With Cerebrovascular Accident; Randomized Controlled Trial
Brief Title: Effect of Mendelsohn Maneuver, Effortful Swallow Training, and the Shaker Exercise on Swallowing Ability Among Dysphagic Patients With Cerebrovascular Accident
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Shahlaa Ali, PhD student, Adult Nursing Department, Principal Investigator, nurse, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dysphagic Patients with CVA
Record Dates: First submitted 2025-09-25; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Neurogenic Dysphagia

STUDY DESIGN:
Intervention Model Description: Research design: True-experimental research design will be used to investigate the effect of the swallowing exercises on improving the post stroke dysphagia. This study used to estimate the effect of an intervention on its target population with randomization .
  * The sample groups must be assigned randomly.
  * There must be a viable control group.
  * Only one variable can be manipulated and tested.
  * The tested subjects must be randomly assigned to either control or experimental groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mendelsohn maneuver (Other): Mendelssohn's First, the participant was given a tiny quantity of food or liquid in their mouth. In cases where there was a possibility of aspiration, dry swallowing was employed. Second, the thumb and fingers were used to hold the thyroid gland's cartilage. Thirdly, the dry swallowing technique was mandated by the subject therapist. Fourth, as the patient swallows, the thyroid cartilage is pulled upward. Fifth, the patient should hold the thyroid cartilage at its highest moveabl position for two seconds. Sixth, the person should be at ease. Seventh, go through steps 1 through 6 again, 15 to 20 times.
  Interventions: Other: Compare the effect of Mendelsohn maneuver, effortful swallow training, and the Shaker exercise on neurogenic dysphagia among stroke patients.
- Effortful Swallow (Other): Effortful Swallow: Patients will be instructed to squeeze hard with all of their tongue muscles when they swallow. This technique will be performed twice daily, in the morning and in the evening for five consecutive days. Dysphagia exercises will be carried out five days a week for two weeks.
  Interventions: Other: Compare the effect of Mendelsohn maneuver, effortful swallow training, and the Shaker exercise on neurogenic dysphagia among stroke patients.
- Shaker Exercise (Other): Shaker Exercise : Patients will be taught to lie in a recumbent position, look at their toes, and raise their head without lifting their shoulders toward their chest. They maintain this posture for a minute before taking a brief break and repeating the head-raising motion. For five days in a row, the exercise will performed twice a day in the morning and the afternoon. Dysphagia exercises will be carried out five days a week for two weeks.
  Interventions: Other: Compare the effect of Mendelsohn maneuver, effortful swallow training, and the Shaker exercise on neurogenic dysphagia among stroke patients.

INTERVENTIONS:
Other: Compare the effect of Mendelsohn maneuver, effortful swallow training, and the Shaker exercise on neurogenic dysphagia among stroke patients. — To achieve single blind in this trial, the participant is kept blinded to their group assignment (interventions and control groups) throughout the study. The data collector administers the assigned intervention (Mendelsohn maneuver, effortful swallow training, and the Shaker exercise ) without revealing the participant's group assignment. The researcher retains knowledge of group allocation to ensure Single blind. Interventions are randomized, and assess Effect of Mendelsohn maneuver, effortful swallow training, and the Shaker exercise on swallowing Ability without knowing the type of maneuvers received, ensuring that participants' expectations do not influence the results. These procedures reduce the influence of prior expectations and ensure an effective study.

SUMMARY:
The study aims to Compare the effect of Mendelsohn maneuver, effortful swallow training, and the Shaker exercise on neurogenic dysphagia among stroke patients.

DETAILED DESCRIPTION:
Stroke is a significant global challenge for healthcare personnel, as it is a leading cause of disability and death globally. (1) There are two primary categories of stroke: ischemic and hemorrhagic. Stroke results in functional disabilities, with 15-30% of individuals experiencing persistent impairments for the duration of their lives. (2) Stroke is the foremost life-threatening and significant neurological ailment that causes disability, According to predictions from the World Health Organization (WHO), strokes will become the second most common cause of death, behind ischemic heart disease, in both developed and developing nations by 2020. (3) From a clinical standpoint, stroke occurs when the blood flow to the brain is interrupted due to either a blockage in the main blood vessels produced by thromboembolism or the bursting of arteries. The majority of strokes, over 85%, are ischemic in nature, resulting from the obstruction of brain arteries due to thrombotic or embolic occlusion. (4) Neurogenic Dysphagia is a condition where the complex and integrated sensory system is impaired. It commonly affects individuals with various neurological diseases, particularly acute stroke. (5) Dysphagia, in fact, is a highly perilous outcome of stroke that can result in lung infections and even mortality among stroke patients. Hence, it is important to conduct accurate screening, diagnosis, and treatment of dysphagia in patients with acute stroke in order to enhance their quality of life and perhaps mitigate the risk of mortality. (6)

ELIGIBILITY:
Inclusion criteria:

1. An adult patient diagnosed with stroke.
2. Patients who had been diagnosed with dysphagia after stroke.
3. Patients who are hemodynamically stable, conscious and have adequate cognitive ability to follow simple instructions and able to sit upright for at least 30 minutes.

Exclusion criteria:

1. Unstable angina and myocardial infarction)MI(.
2. History of seizure.
3. Head injury or neurological disease other than stroke, neurosurgery .
4. Oral and maxillofacial surgery.
5. Dysphagia prior to stroke.
6. Gastrointestinal tract upsets.
7. Patients who receive hypnotics or sedation.
8. critical ill.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Gugging swallowing screen | The data collection period 12 weeks
  Gugging Screen: The instrument focuses on the swallowing screen (guss) developed by Michaela Trapl et al. 2007, S, which will be used to assess the severity of dysphagia in participants. The English version will be used.Two component are involved in the GUSS that's are: part 1 (indirect swallow test) also called the preliminary assessment, and part 2 (the direct swallow test). A point system was chosen, with a maximum of five points that can be scored in each subtest, where higher numbers indicate healthier performance. To move on to the next subtest, you have to reach this maximum. Every test item has a value of either one point (physiologic) or zero points (pathologic). We employed a new rating inside the direct swallowing test's scoring criteria for "deglutition." Pathologic swallowing receives 0 points, delayed swallowing receives 1 point, and normal deglutition receives 2 points. To receive the maximum score of five points on the subtest.

CONTACTS AND LOCATIONS:
Overall Officials: shahlaa Ali, Study Director — Baghdad University

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.